CLINICAL TRIAL: NCT04228328
Title: Validity and Reliability of the 6-minute Walk Test Over a Distance of 6 Metres in People With Multiple Sclerosis
Acronym: VR6minWT6
Status: Completed | Type: Observational
Sponsor: Haute Ecole de Santé Vaud (Other)
Collaborators: University of Applied Sciences of Western Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-01864
Record Dates: First submitted 2020-01-10; First posted 2020-01-14 (Actual); Results first posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Walk Test

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: The 6-minutes Walk Test — To walk for 6 minutes

SUMMARY:
The objective of this study is to validate a different version of the 6 minutes Walk Test (6minWT), the 6minWT on 6 meters, instead of the 30 meters.

The secondary objectives are to verify the reliability of this new version and to analyze the possible differences between the 6minWT6 and the 6minWT30 (according to speed at half-turn, other parameters: age, gender, height, EDSS score, type of disease, time since relapse).

DETAILED DESCRIPTION:
The 6minWT is used by physiotherapists to monitor the walking endurance abilities of multiple sclerosis (MS) patients. The protocol for this test recommends a distance of 30 meters (6minWT30) to perform the test. However, this distance is not always available in practices and patients' homes. The aim of this study is therefore to validate a protocol over a distance of 6 meters (6minWT6) and to evaluate its reliability : intra-evaluator and test-retest.

The project focuses on the population of walking patients with MS. Inclusion: adults, confirmed diagnosis of MS, Expanded Disability Status Scale (EDSS) score 3 to 6.5, or be able to walk 30 metres with or without aids, good understanding of French, have already completed a 6-minute walking test, be able to give consent by signature.

Exclusion: Lung disease, heart disease, co-morbidity preventing 6minWT, relapse in the last 3 months, chronic fatigue ≥ at 8 (Visual Analog Score-Fatigue or Rochester Fatigue Diary).

21 participants will be needed to obtain a good correlation coefficient, which is the objective of the validation of the new version of the 6minWT. The alpha was set at 0.01, the power at 0.9 for a correlation of 0.8.

Each patient will enter the study for one week, corresponding to two visits. The participant will perform the 6minWT6 and the 360 Degree Turn Test the first day and the 6minWT30 followed by the 6minWT6 after up to 45 minutes rest, the second day, a week apart.

ELIGIBILITY:
Inclusion Criteria:

* adults
* confirmed diagnosis of MS
* Expanded Disability Status Scale score 3 to 6.5 or to be able to walk 30 meters with or without aids
* good understanding of French
* have already completed a 6-minute walk test
* to be able to give consent by signature

Exclusion Criteria:

* Lung disease
* Heart disease
* co-morbidity preventing 6minWT
* relapse in the last 3 months
* chronic fatigue ≥ at 8 (Visual Analog Scale- Fatigue)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Multiple sclerosis patient able to walk at least 30 meters, Expanded Disability Status Scale from 3 to 6.5
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2020-11-05 (Actual); Study Completion 2020-11-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenny Guex, PhD, Principal Investigator — Haute Ecole de Santé Vaud
Locations (1):
- Haute Ecole de Santé Vaud, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: On 32 patients pre-screened, 4 could not be reached by phone, 1 left for another country, 1 suffered too much from heath, 4 did not met inclusion criteria and 1 finally withdrew : 21 were enrolled
Groups:
- Test Group: Participants walked for 6 minutes on a 6-m walkway, did the 360 Degree Turn Test, walked for 6 minutes on a 30-m walkway and again a 6 m walkway.
Period: Overall Study
Arm/Group | Test Group
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Test Group: Participants walked for 6 minutes on a 6-m walkway, did the 360 Degree Turn Test, walked for 6 minutes on a 30-m walkway and again a 6-m walkway.
Arm/Group | Test Group
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  Switzerland | 21
Height [Mean (Standard Deviation); unit: cm] | 168 (5.6)
Weight [Mean (Standard Deviation); unit: kg] | 64 (10)
Type of MS [Count of Participants; unit: Participants]
  Relapsing-remitting | 10
  Secondary progressive | 10
  Primary progressive | 1
Expanded Disability Status Scale [Median (Inter-Quartile Range); unit: units on a scale] — The Expanded Disability Status Scale (EDSS) is a scale aimed to quantifying disability in multiple sclerosis. The EDSS scale ranges from 0 to 10 in 0.5 unit increments. 10 is the highest level of the scale and represent death. From 0 to 3.5, people are able to walk without aid. From 3.5-6.5, people are defined by the impairment to walking. From 7, people are dependant and restricted to wheelchair or bedridden. Scoring is based on an examination by a neurologist. It was collected through the participant or direct contact with their neurologist.
  units on a scale | 4.75 [3.75 to 6.0]
Disease duration [Median (Inter-Quartile Range); unit: years] | 19 [14 to 31]
Assistive device [Count of Participants; unit: Participants]
  None | 9
  1 crutch | 2
  2 walking sticks | 4
  2 crutches | 1
  Walker | 5
Time since last relapse [Median (Inter-Quartile Range); unit: month] | 60 [30 to 108]
Medication [Count of Participants; unit: Participants]
  None | 10
  Interferon | 2
  Fingolimod | 1
  Ocrelizumab | 8
Visual Analogue Scale for Fatigue [Median (Inter-Quartile Range); unit: units on a scale] — The Visual Analogue Scale for Fatigue is aimed to easily and quickly quantify the level of fatigue. The participant had to stick his current level of fatigue on a blank line of 10 cm where "extreme fatigue" was mentioned to the right and "no fatigue" to the left. A corresponding graduated line allowed the tester to transform the sticked level of fatigue in a unit between 0 (no fatigue) to 10 (extreme fatigue).
  units on a scale | 2 [1 to 3]
Regular physical activity [Median (Inter-Quartile Range); unit: min] | 90 [50 to 130]

OUTCOME MEASURES:

1. Primary Outcome: The 6-minutes Walk Test on 6 Meters
Description: The patient walk for 6 minutes back and forth in a 6-meter hallway turning around cones.
Time Frame: First test day
Measure: Mean (Standard Deviation); unit: m
Groups:
- Test Group: Participants walked for 6 minutes on a 6 m distance, did the 360 Degree Turn Test, walked for 6 minutes on a 30 m distance and again a 6 m distance.
Arm/Group | Test Group
Number analyzed (Participants) | 21
m
  Tester measured | 215.86 (113.8)
  Video-verified | 221.57 (113.8)

2. Secondary Outcome: 360 Degree Turn Test (Time)
Description: The person must complete a full lap on himself or herself and the execution time is measured
Time Frame: First test day
Measure: Mean (Standard Deviation); unit: s
Arm/Group | Test Group
Number analyzed (Participants) | 21
s | 6.00 (4.11)

3. Secondary Outcome: 360 Degree Turn Test (Number of Steps)
Description: The person must complete a full lap on himself or herself and the number of steps is measured
Time Frame: First test day
Measure: Mean (Standard Deviation); unit: number of steps
Arm/Group | Test Group
Number analyzed (Participants) | 21
number of steps | 8.16 (3.59)

4. Secondary Outcome: 6 Minute Walk Test on 30 Meters
Description: The patient walk for 6 minutes back and forth in a 30-meter hallway turning around cones.
Time Frame: Second test day
Measure: Mean (Standard Deviation); unit: m
Arm/Group | Test Group
Number analyzed (Participants) | 21
m | 295.95 (156.54)

5. Secondary Outcome: The 6-minutes Walk Test on 6 Meters
Description: The patient walk for 6 minutes back and forth in a 6-meter hallway turning around cones.
Time Frame: Second test day
Measure: Mean (Standard Deviation); unit: s
Arm/Group | Test Group
Number analyzed (Participants) | 21
s
  Tester measured | 227.05 (123.49)
  Video-verified | 228.90 (122.87)

ADVERSE EVENTS:
Time Frame: 1 week
Description: no adverse event to be reported
Groups:
- Test Group: Participants walked for 6 minutes on a 6-m walkway, did the 360 Degree Turn Test and walked for 6 minutes on a 30-m walkway and again a 6-m walkway.
Arm/Group | Test Group
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-10): https://cdn.clinicaltrials.gov/large-docs/28/NCT04228328/Prot_SAP_000.pdf